CLINICAL TRIAL: NCT03429868
Title: Prognostic Value of the Integrated PET/MRI in Patients With Nasopharyngeal Carcinoma
Brief Title: PET and MRI in Prognosis Prediction of NPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NSC 104-2314-B-182A-084-MY3
Record Dates: First submitted 2018-02-06; First posted 2018-02-12 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2020-05

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; Nead neck cancer; Prognosis; PET; MRI
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- integrated PET/MRI (Experimental): The participants receive an integrated 18F-FDG PET/MRI during tumor staging.
  Interventions: Device: integrated PET/MRI

INTERVENTIONS:
Device: integrated PET/MRI — The participants receive an integrated 18F-FDG PET/MRI scan in addition to the conventional 18F-FDG PET/CT on the same day during tumor staging.
  Whole body 18F-FDG PET/CT is performed one hour after injection of 10mCi of 18F-FDG. 18F-FDG PET/MRI is done after the PET/CT scan. And no additional 18F-FDG is given to the patients in the PET/MRI scan.

SUMMARY:
Nasopharyngeal carcinoma (NPC) differs from other head and neck malignancies terms of its epidemiology, pathology, and treatment outcome. Integrated PET/MRI is a new imaging modality, which can simultaneously acquire PET and MRI images. Considering the lack of reports on the use of hybrid PET/MRI systems in prognosis prediction in NPC, the investigators conduct this prospective study to investigate the roles of integrated PET/MRI parameters for predicting treatment outcome and prognosis in patients with NPC.

DETAILED DESCRIPTION:
1. Background:

   Nasopharyngeal carcinoma (NPC) has a higher local tumor control rate but a higher incidence of distant metastasis compared with squamous cell carcinomas of other regions of the head and neck. Thus, it's usually considered a distinct study group. A reliable clinical prognostic factor for NPC patients is still lacking. Positron emission tomography (PET) with 2- [fluorine- 18]fluoro-2-deoxy-D-glucose (18F-FDG)/computed tomography (CT) has been used extensively for diagnosis and assessment of prognosis in NPC in recent years. Several PET-derived imaging parameters such as standardized uptake value (SUV), metabolic tumor volume (MTV), or total lesion glycolysis (TLG) have been proposed as potential prognosticators in NPC. MRI functional parameters also play a role to assess the cellular or molecular change of head and neck cancer. Diffusion-weighted MR imaging (DWI) is a technique, which can quantify the diffusion of water molecules in tissues using apparent diffusion coefficient (ADC). ADC is inversely correlated with cellular density. Dynamic contrast-enhanced perfusion MR imaging (DCE-MRI) is another MRI technique based on sequential imaging obtained during the passage of a contrast of agent through the tissue. It enables probing the microvascular environment in the tumor tissue.

   Integrated PET/MRI is a new imaging modality, which can simultaneously acquire PET and MRI images. Traditionally, PET and MRI images were acquired on different dates and were fused by commercial software. Problems caused by a separate system include SUV or MRI parameters were reported to be different if the scans were acquired on different days. Simultaneous acquisition of PET and MRI images would solve these problems.
2. Aim: The investigators conduct this prospective study to investigate the roles of integrated PET/MRI imaging parameters for predicting treatment outcomes and prognosis in patients with NPC.
3. Study design:

Patients: All patients receive whole-body 18F-FDG PET/MRI following 18F-FDG-PET/CT on the same day. For tumor staging, the 7th edition of the American Joint Committee on Cancer (AJCC)/Union for International Cancer Control (UICC) cancer staging system is used. The patients with stage I disease are treated with definitive radiation therapy alone, while patients with stage II-IVB are treated with concurrent chemoradiotherapy. Patients with metastatic disease (stage IVC) are treated with standard platinum-based chemotherapy.

18F-FDG PET/CT: All study patients fast for at least 6 h before 18F-FDG PET/CT imaging. Scans are performed using a Biograph mCT scanner (Siemens Medical Solutions, Malvern, PA, USA) consisting of a four-ring PET scanner (axial field-of-view [FOV] = 22.1 cm, transaxial FOV = 70 cm) and a 40-section CT scanner.

Whole-body 18F-FDG PET/MRI: PET/MRI is performed on a Biograph mMR (Siemens Healthcare, Erlangen, Germany) following the PET/CT scan on the same day. The PET/MRI system is equipped with 3-T magnetic field strength, total imaging matrix coil technology covering the entire body with multiple integrated radiofrequency surface coils, and a fully functional PET system with avalanche photodiode technology embedded in the magnetic resonance gantry.

Image interpretation: The PET/CT and PET/MRI data sets are evaluated on dedicated workstations (Syngo.via, Siemens Healthcare, Erlangen, Germany). The readers interpret the (1) MR images from PET/MRI, (2) 18F-FDG PET/MRI images, and (3) 18F-FDG PET/CT images independently. They are aware of the study protocol but are blinded to the results from the other imaging modalities. Imaging parameters including SUV, MTV, TLG, ADC, Ktrans, Ve, and Vp are calculated.

Statistical analysis: Overall survival (OS) and recurrence-free survival (RFS) serves as the main outcome measures. OS is calculated from the date of diagnosis to the date of death or censored at the date of the last follow-up for surviving patients. RFS is defined as the time between the end of treatment and the date of recurrence (tumor relapse or death) or censored at the date of the last follow-up. The cutoff values for the clinical variables and imaging parameters in survival analysis are determined using the log-rank test based on the RFS and OS rates observed in the entire study cohort. Survival curves are plotted using the Kaplan-Meier method. The effect of each individual variable is initially evaluated using univariate analysis. Cox regression models are used to identify the predictors of survival. Two-tailed P values < 0.05 are considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven primary nasopharyngeal carcinoma
2. Age > or = 20
3. Willing to receive therapy
4. The ability to provide written informed consent and receive the scheduled scans

Exclusion Criteria:

1. Woman with pregnancy or during lactation
2. A history of other malignancies or concomitant cancers in different anatomical locations
3. Not suitable to receive the PET scan such as serum glucose levels of > 200 mg/dL or space phobia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years
  Being calculated from the date of diagnosis to the date of death or censor at the date of the last follow- up for surviving patients.

SECONDARY OUTCOMES:
Recurrence-free survival | 3 years
  The time between the end of treatment and the date of recurrence (tumor relapse or death) or censor at the date of the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Chieh Chan, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan SC, Ng SH, Yeh CH, Lin YC, Lin CY, Wang JH, Cheng NM, Chen SH, Chang KP, Hsieh JC. Prognostic utility of 18F-FDG PET/MRI with intravoxel incoherent motion imaging in nasopharyngeal carcinoma. Eur J Nucl Med Mol Imaging. 2025 Dec;53(1):338-349. doi: 10.1007/s00259-025-07425-6. Epub 2025 Jul 2. PMID 40601020